CLINICAL TRIAL: NCT04351633
Title: Psychological Impact of Quarantine in Osteoporosis Patient During COVID-19 Outbreak
Acronym: OsPsyCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_31; 2020-A00911-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2; Osteoporosis
Keywords: Psychological impact; COVID-19
MeSH Terms: conditions — Osteoporosis; COVID-19

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- osteoporosis patient
  Interventions: Other: questionnaire assesment

INTERVENTIONS:
Other: questionnaire assesment — questionnaire assesment

SUMMARY:
In the context of quarantine with COVID-19, we wish to study the experience and psychological impact in adult patients living with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with osteoporosis
* Patient in confinement
* Patient with sufficient understanding of the French language

Exclusion Criteria:

* Non adult patient
* patient without quarantine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: osteoporosis patient will be interviewed par internet questionnaire (patient association / AFLAR)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
percentage of patient with feeling of disabilities | maximum 1 week from baseline on

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cortet, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France